CLINICAL TRIAL: NCT03178604
Title: Comparison Between Classic and Sham Massage on Psychological and Physical Functional Variables in Athletes: A Randomized Pilot-Placebo Trial.
Brief Title: Classic and Sham Massage on Psychological and Physical Functional Variables in Athletes
Acronym: MHams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Dr, University of Valencia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ID0015
Record Dates: First submitted 2017-06-03; First posted 2017-06-07 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Hamstring Contractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic massage (Active Comparator): Classic massage (CM) treatment based on petrissage. It applies: 1 minute of mild effleurage, 5 minutes of deep effleurage with the thumbs, 5 minutes of firm kneading and 1 minute of tapotement (20 minutes in total). This procedure was repeated for each muscle group.
  Interventions: Other: Classic massage
- Sham massage (Active Comparator): Sham massage (SM). 20 minutes in total soft effleurage was performed. This procedure was repeated for each muscle group.
  Interventions: Other: Sham massage

INTERVENTIONS:
Other: Classic massage — It involves applying the classic massage techniques: effleurage (gliding or sliding movement over the skin with a smooth continuous motion following the direction of the muscle fibers of the superficial muscles in a distal to proximal direction); petrissage (lifting, wringing, or squeezing of soft tissues in a kneading motion, or pressing or rolling of the tissues under or between the hands); tapotement (various parts of the hand striking the tissues at a fairly rapid rate). The general objective is to improve extensibility of muscle, tendon, fascia, joint capsule, and ligamentous structures.
  Arms: Classic massage
Other: Sham massage — This group received a placebo intervention at the same time as the other group, maintaining only soft touch with the participant without exerting any mechanical pressure.
  Arms: Sham massage

SUMMARY:
In this study we intend to apply a treatment protocol for hamstrings that can be beneficial for a good recovery.

Initially, a sample of athletes with hamstring shortening was chosen. Once the sample is chosen, it will be divided into two groups: group 1 (G.1) who will receives a sham massage, group 2 (G.2) that receives the classic massage.

To finalize the study comparing the results of the two groups to observe the experimental protocol obtains better results.

Material and methods The sample of an athletic club. Recruiting subjects between 18 and 45 years old without other injuries of the lower limb. Subjects with shortening of the hamstring muscles are available through the specific shortening test.

This is a randomized controlled trial. Subjects were randomly assigned to two intervention groups (1 treatment and 1 placebo control). The intervention consists of 4 sessions for 1 month. The sessions have a duration of 45 minutes. Evaluations are performed at the beginning of treatment, at the end of treatment. Participants also perform strengthening exercises three days a week, a total of 3 sets with 15 repetitions each.

Group 1 receives a sham massage of the quadriceps and hamstrings. Group 2 receives a classic massage of the quadriceps and hamstrings. The assessments consist of knee and hip goniometry, lumbar and hamstring flexibility by finger-to-floor testing, and complete the questionnaire Mood Status Profile (POMS), Which evaluates the states of mind.

ELIGIBILITY:
Inclusion Criteria:

* The sample comes from two athletic clubs of Valencia with subjects between 18 and 30 years old without lower limb injuries, with shortening of the hamstring muscles selected by the specific shortening test.

Exclusion Criteria:

* Muscle-skeletal injuries in any part of the body are excluded from the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Popliteal test | 4 weeks
  It is a specific test that is performed in supine position. The subject flexes the hip until it reaches 90º, while keeping the knee flexed. Subsequently, he takes the ankle and takes the knee to an extension position passively. In this position, one takes measure of the degrees that are lacking until the complete extension. During the test, it should be ensured that there are no compensations.

SECONDARY OUTCOMES:
Hip flexion test | 4 weeks
  It is performed with a knee and assesses the shortening of the hamstring muscles. The test is performed in supine position, and consists of flexing the hip in a slow and passive way until it reaches a flexion that the tightness or pain that the participant feels does not let go more. It should be noted that there is no knee flexion or any other type of compensation such as tilting of the pelvis. For the quantification we use a universal goniometer.
Range of motion | 4 weeks
  Both legs (hip flexion, knee flexion and knee flexion) are measured by a universal goniometer, which has proven to be a valid and reliable instrument.
Lumbar flexibility | 4 weeks
  By the Fingertip-to-Floor Test (FFT). The restraints placed barefoot on a platform 25 cm high, with feet together and flat and toes on the edge pointing forward. They are then asked to lean forward and try to reach the floor with their fingertips as much as possible without discomfort, keeping the knees and arms fully extended. The bending is maintained for 3 seconds and the vertical distance between the tip of the middle finger and the platform is measured. The best of 3 trials is used for analysis.
Emotional state of the athlete | 4 weeks
  Through the Profile of Mood States Questionnaire (POMS). This scale contains a total of 58 adjectives, which includes 6 dimensions of moods: tension, depression, anger, vigor, fatigue and confusion.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí López, Dr, Principal Investigator — Faculty of Physiotherapy, University of Valencia, Spain
Locations (1):
- Gemma Victoria Espí López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No